CLINICAL TRIAL: NCT03754335
Title: SubArachnoid Hemorrhage HEadache Treated by Lumbar Puncture
Acronym: SAH-HELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RC31/17/0355; 2018-A00629-46 (Other: ID-RCB)
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Headache
Keywords: Aneurysmal subarachnoid hemorrhage; lumbar puncture; headache
MeSH Terms: conditions — Subarachnoid Hemorrhage; Headache | interventions — Spinal Puncture

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, prospective monocentric trial evaluating in parallel groups
Who Masked: Participant, Investigator
Masking Description: This procedure is to be able to easily randomize half of the patients into a "sham" LP arm passed by independent practitioners of the investigators in charge of the patient, which allows a good double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar puncture (Experimental): Lumbar puncture in addition to a predefined analgesic protocol Patients will be randomized between the 3rd and 5th days following aneurismal rupture.
  Interventions: Procedure: Lumbar puncture
- Sham lumbar puncture (Active Comparator): Sham lumbar puncture in addition to a predefined analgesic protocol Patients will be randomized between the 3rd and 5th days following aneurismal rupture.
  Interventions: Procedure: Lumbar puncture

INTERVENTIONS:
Procedure: Lumbar puncture — Patient will be managed according to the current international recommendations in the Toulouse acute stroke center.
  In the absence of clear recommendation in the literature headache will be treated according to our local predefined analgesic protocol: paracetamol 1g/6 h, and if the numerical scale ≥ 4 : continuous intravenous morphine starting at 1mg/h and increased per 0.5 mg/h every hour if numerical scale remains ≥ 4.
  Lumbar puncture will be performed between day 3 and day 5 after subarachnoid hemorrhage onset by an independent scientist from our clinical investigator center. 30-mL CSF will be removed by LP.
  Sham LP consisting in superficial skin puncture by a subcutaneous needle (27 gauge needle) during the usual procedure will be performed at the same time point.
  Other Names: Sham Lumbar Puncture

SUMMARY:
Headache control is one of the major challenges in patients who suffered an acute aneurysmal subarachnoid hemorrhage (aSAH). Headache affects 90% of the patient and is resistant to the major pain medication. It results from the increased intracranial pressure and the inflammation caused by the accumulation of arterial blood in the subarachnoid space. Hemorrhagic cerebrospinal fluid (CSF) removal by a lumbar puncture (LP), is well tolerated, reduces intracranial pressure and accelerates the clearance of the blood products from CSF. Nonetheless it has never been tested in a randomized trial. The investigators aim to compare in patients who experienced a low grade aSAH, the variation of headache intensity after CSF removal by LP vs. Sham LP in addition to predefined analgesic protocol management.

DETAILED DESCRIPTION:
After aneurysmal subarachnoid hemorrhage (aSAH) almost 90 % of patients experience a severe headache during their hospital stay. Pain control often requires high doses of opioid drugs and sedation that remain only partially efficacious. In addition, there is to the investigator's knowledge currently no recommendation or consensus on aSAH related headache management. aSAH related headache results from the prolonged increased intracranial pressure and meningeal inflammation related to the accumulation of blood products in the subarachnoid space. Preliminary studies, suggest that hemorrhagic cerebrospinal fluid (CSF) removal by lumbar puncture (LP) or lumbar drain, is safe and decreases intracranial pressure. However its impact on headache control has never been tested. A reliable headache evaluation has to be performed among conscious patients experiencing a "low-grade" aSAH.

The objective of the study is to evaluate in patients experiencing low-grade acute aSAH (WFNS 1-3), the efficacy of CSF removal by LP vs. sham LP, on headache control. 74 patients with secured aneurysm by coiling, will be randomized (1:1) between day 3 and day 5 after aneurysmal rupture. The procedure will be performed in addition to a pre-specified antalgic protocol.

Mean headache intensity will be measured with the numeric verbal scale during the 24 hours before and the 24 hours after the procedure. The variation of mean intensity will be compared between the 2 groups.

The investigators hypothesize that this treatment may significantly decrease headache intensity after an aSAH. If this hypothesis is confirmed CSF removal by LP could be a simple cost effective and worldwide available strategy to improve

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Low grade subarachnoid hemorrhage (WFNS score between 1 and 3)
* Aneurysmal rupture ≤ 5 days
* Ruptured aneurysm secured by coiling since at least 48 h
* Headache with a mean numeric verbal scale ≥ 4/10 during the last 24 hours
* No contraindication for lumbar puncture
* Affiliation to french social security
* Person able to express her consent and to assess own headache intensity

Exclusion Criteria:

* Minor,
* Pregnancy, breastfeeding
* Subarachnoid hemorrhage without aneurysm
* Ruptured aneurysm not secured
* High grade (WFNS 4 and 5) subarachnoid hemorrhage
* Efficient anticoagulation
* External ventricular drain placed before randomisation
* People under legal protection
* Participation to another research study with an ongoing disqualification period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Difference of headache mean intensity variation measured after a lumbar puncture or a sham LP. | 24 hours after the inclusion
  The mean intensity will be assessed using the verbal rating scales (VRS). It is a scale administered by the medical team, which brings together the score given by the patient between 0 and 10 (0 = absence of pain; 10 = maximum of conceivable pain)Headache mean intensity variation will be calculated by the difference between these scores evaluated 24 hours before and the 24 hours after the procedure.

SECONDARY OUTCOMES:
Difference of variation in the mean intensity of headache | 48 hours
  Difference of variation in the mean intensity of headache measured by the nurse in charge of the patients every 4 h between the 24 hours before and the 24 hours after the procedure. Difference of variation will be assessed using the verbal rating scales (VRS). It is a scale administered by the medical team, which brings together the score given by the patient between 0 and 10 (0 = absence of pain; 10 = maximum of conceivable pain). Headache mean intensity variation will be calculated by the difference between these scores evaluated 24 hours before and the 24 hours after the procedure.
Difference of maximal headache intensity | 48 hours
  Difference of maximal headache intensity will be assessed using the verbal rating scales (VRS). It is a scale administered by the medical team, which brings together the score given by the patient between 0 and 10 (0 = absence of pain; 10 = maximum of conceivable pain). Headache maximal intensity variation will be calculated by the difference of maximal headache intensity measured during 24 hours before and 24 hours after the procedure by the nurse in charge of the patients every 4 hours.
Kinetic of headache intensity | 7 days
  Kinetic of headache intensity during the 7 days following the procedure (global assesment by the patient and mean/max of measurement every 4 hours). The headache intensity will be assessed using the verbal rating scales (VRS). It is a scale administered by the medical team, which brings together the score given by the patient between 0 and 10 (0 = absence of pain; 10 = maximum of conceivable pain).
Difference of responding patients | 7 days
  Difference of responding patients defined by patients with a decreased of the mean intensity of 30 % and 50 %, 24 hours after the procedure and daily during the 7 days following the procedure.
Occurrence of a clinical deterioration | 1 day
  Related to the other complication of subarachnoid hemorrhage : Occurrence of a clinical deterioration related to delayed cerebral ischemia assessed by NIHSS and GCS) and the occurrence of a new infarction on follow-up MRI.
Persistence of Chronic hydrocephalus | 3 month
  Rate of chronic hydrocephalus defined by the modification of the ventricle size between the post interventional MRI and the follow-up MRI at 3 months.
Improvement of the clinical global impression | 3 months
  Disability and Quality of life : Improvement of the "Clinical Global Impression -Improvement" (CGI-I) at 24 hours, day 7 and 3 months (clinical improvement defined by a score of 1 or 2). The CGI-I is used by clinicians to rate improvement in a subject's condition (benefits) since baseline. It is a 7-point scale with 1=very much improved, 2=much improved, 3=minimally improved, 4=not changed, 5=minimally worse, 6=much worse; and 7=very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Calvière, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No